CLINICAL TRIAL: NCT01670773
Title: A Phase 1, Single Center, Biomarker Study in Healthy Subjects Receiving Single Doses of CAT-1004
Brief Title: A Study of CAT-1004 Biomarkers in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Catabasis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: CAT-1004-103
Record Dates: First submitted 2012-08-16; First posted 2012-08-22 (Estimated); Last update posted 2012-10-30 (Estimated); Status verified 2012-10

CONDITIONS: Assessment of Mechanistic Blood Biomarkers in Healthy Humans
MeSH Terms: interventions — edasalonexent; salicylsalicylic acid

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- CAT-1004 Dose #1 (Experimental): Single dose #1
  Interventions: Drug: CAT-1004
- Salsalate + DHA (Active Comparator): Single dose #2
  Interventions: Drug: Salsalate + DHA
- Placebo (Placebo Comparator): Single Dose #3
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CAT-1004
  Arms: CAT-1004 Dose #1
Drug: Salsalate + DHA
  Arms: Salsalate + DHA
Drug: Placebo
  Arms: Placebo

SUMMARY:
This study is being conducted to assess mechanistic blood biomarkers of CAT-1004 in healthy humans.

ELIGIBILITY:
Inclusion Criteria:

* Good health as determined by medical history, vital signs, EGC, physical exam and clinical lab results
* BMI between 18 and 30 kg/m2 inclusive

Exclusion Criteria:

* Viral or bacterial infection within 21 days prior to randomization
* Use of prescription drugs, nonprescription drugs, herbals and dietary supplements within 7 days prior to randomization

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2012-08; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Change in nuclear factor kappa-light-chain-enhancer of activated B cells (NF-kB) activity p65 following ex vivo lipopolysaccharide stimulation | Pre/post each of 3 Single doses

OTHER OUTCOMES:
Other biomarkers including select cytokines and RNA gene expression may also be assessed | Pre/post each of 3 Single doses

CONTACTS AND LOCATIONS:
Overall Officials: Joanne Donovan, MD, PhD, Study Director — Catabasis
Locations (1):
- ProMedica, Brighton, Massachusetts, United States